CLINICAL TRIAL: NCT03324633
Title: Inter Cohorts and Clinical Centres Collaborations of Subjects Co-infected With Hepatitis C and Human Immunodeficiency Virus (Collaboration Inter Cohortes et Centres Cliniques de Sujets Co-infectés Par Les Virus de l'immunodéficence Humaine et de l'hépatite C)
Brief Title: Inter Cohorts and Clinical Centres Collaborations of Subjects Co-infected With HIV and HCV
Acronym: CO13Hepavih
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Bristol-Myers Squibb (Industry); GlaxoSmithKline (Industry); Merck Serono International SA (Industry); Roche Pharma AG (Industry); Schering-Plough (Industry)
Responsible Party: Sponsor
Other Study IDs: ANRS CO13 Hepavih cohort
Record Dates: First submitted 2017-03-21; First posted 2017-10-30 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: HIV; Hepatitis C
Keywords: HIV; HCV; cohort; natural history; cure
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The ANRS CO13 HEPAVIH cohort is a prospective and multicentric cohort created in 2005 with the originality to cover two therapeutic domains of key importance, AIDS and hepatitis C. The cohort, is unique in Europe with more than 1800 participants followed over 10 years including quality of life and compliance to treatment data.

DETAILED DESCRIPTION:
The cohort has been created in 2005 with the general objective to better define the natural history of HCV/HIV co-infection in terms of morbidity and mortality. Furthermore, the cohort aims to determine factors associated with morbidity and mortality and to better understand interactions between the two viruses and their respective treatments.

The ANRS CO13 Hepavih is currently composed of 28 french metropolitan clinical centers of infectious diseases and hepatogy diseases (mostly teaching hospital).

The period of patient inclusion has been divided in three distinct phases: the first phase (Phase 1) that started in 2005 and ended in 2008, was dedicated to the inclusion of adult HCV/HIV co-infected patients. The following inclusion phase (Phase 2) that concerns patients who received a triple-agent anti-HCV therapy including Boceprevir or Telaprevir, started in 2008 and ended in march 2016. The third one (Phase 3) focusing on patients initiating a DAA anti HCV treatment started in June 2014 and ended in November 2015. Regarding Phase 3, the specific objectives were organized into five thematic domains including clinic, virology, pharmacology, public health and methodology.

Since 31 march 2016, the inclusions are closed and 1,850 patients have been included. The ended of the follow-up is planned on the 31 december 2018.

At the inclusion and during the follow-up period (at least once a year or every 6 months in case of cirrhosis, until 2018 and probably also beyond that date), each HCV/HIV co-infected patient is offered a clinical examination as well as an interview. Additional self-questionnaires are filled by the included patients at the same time points (Social sciences data). The types of data collected from each co-infected patient included in the cohort are organized according to five major thematic classes: socio-demography and behavior, HIV characteristics, HCV characteristics, clinical relevant events, anthropometry, paraclinic data.

The ANRS CO13 HEPAVIH cohort has the purpose to become a facility for specific research regarding the physiopathological and therapeutic aspects of the HCV/HIV co-infection at the disposal of the entire scientific community.

In july 2016, the cohort has pusblished 29 originals articles and 10 as a part of national and European collaborations.

The ANRS CO13 HEPAVIH cohort has adopted functional governance. The Steering Committee, made-up of clinicians, methodologist, the sponsor as well as the cohort coordinators, is focused on logistic and operational aspects of the cohort. The Scientific Committee is the scientific decision-making organization, made-up with scientist experts in main research fields including methodology, hepathology, infectiology, pharmacology, virology and social science, and representatives of the ANRS and patient organizations. It assesses requests for the access to the cohort and provides advices on scientific, methodological and ethical aspects in order to ensure an effective scientific conduct of the research. The Steering Comitee meet once a month and the Scientific Comitee 2/3 times a year.

ELIGIBILITY:
Inclusion Criteria:

All phases of inclusion:

* Patients aged ≥18 years,
* Cover by a social security,
* Able to understand the consent conform.

Phase 1:

* HIV-1/HCV chronically infected (positive HIV antibody test, and HCV RNA positive at inception or negative after anti-HCV treatment)

Phase 2:

* HIV-1/HCV chronically infected (positive HIV antibody test, and HCV RNA positive at inception or negative after anti-HCV treatment) treated with protease inhibitor based treatment (PegIFN, Ribavirin and Telaprevir or Boceprevir) or having cleared HCV spontaneously in the absence of anti-HCV treatment

Phase 3:

* HIV-1/HCV chronically infected (positive HIV antibody test, and HCV RNA positive at inception or negative after anti-HCV treatment) treated with DAA anti-HCV treatment (all combinations)

Exclusion Criteria:

* Patients <18 years old
* So-called vulnerable populations (minors, people under guardianship or protection, or a private individual under protection from making legal or administrative decisions)
* Without an healthcare insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Co-infected patients with HIV and HVC who are usually treated in one of the clinical centres of the ANRS CO13 Hepavih network (28 located in metropolitan France since 2014)
Sampling Method: Non-Probability Sample
Enrollment: 1850 (Actual)
Dates: Start 2005-06; Primary Completion 2017-09 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Improve effectiveness and quality of medical care in Hepatitis C in HIV patients | Through study completion : One visit/year for each participant + one additionnal visit every 6 months for patients with a cirhhosis
  The CRFs compile clinical, biological, genetic and virological data : Clinical events, treatments (HIV, HVC, others), clinical exams (height, weight, hip and waist circumferences), virological : CD4, CD8, HIV RNA, HVC RNA (+genotype), HVB serology, liver functions tests and biology (fibroscan, fibrotest, ultrasound, transaminases, bilirubin, alkaline phosphatase, gamma GT,...), metabolic biochemistry (glycemia, insulin, cholesterol, creatinin, lipase). Patients also completed sociales sciences questionnaires (quality of life, depression,...) During the annual visit, samples are taken : blood for DNA, serum and plasma and are stocked in a biobank used for scientific projects.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Salmon, MDPhD, Principal Investigator — Assistance Publique des Hôpitaux de Paris -Université Paris Descartes; Linda Wittkop, MDPhD, Principal Investigator — Inserm U1219 CHU de Bordeaux-Université de Bordeaux

IPD SHARING:
Plan to Share IPD: Yes
Data have been already shared in context of national, european and international collaborations : ANRS CO12 CIRVIR, ANRS HC EP25 PRETHEVIC, DHOS FIBROSTIC COHERE, … and also with industrial partners.

REFERENCES:
- [Result] Sogni P, Gilbert C, Lacombe K, Piroth L, Rosenthal E, Miailhes P, Gervais A, Esterle L, Chas J, Poizot-Martin I, Dominguez S, Simon A, Morlat P, Neau D, Zucman D, Bouchaud O, Lascoux-Combe C, Bani-Sadr F, Alric L, Goujard C, Vittecoq D, Billaud E, Aumaitre H, Boue F, Valantin MA, Dabis F, Salmon D, Wittkop L. All-oral Direct-acting Antiviral Regimens in HIV/Hepatitis C Virus-coinfected Patients With Cirrhosis Are Efficient and Safe: Real-life Results From the Prospective ANRS CO13-HEPAVIH Cohort. Clin Infect Dis. 2016 Sep 15;63(6):763-770. doi: 10.1093/cid/ciw379. Epub 2016 Jun 17. PMID 27317796
- [Result] Marcellin F, Protopopescu C, Poizot-Martin I, Miailhes P, Esterle L, Wittkop L, Spire B, Bocquier A, Salmon-Ceron D, Dabis F, Carrieri MP; HEPAVIH ANRS CO13 Study Group. Short article: Fatigue in the long term after HCV treatment in HIV-HCV-coinfected patients: functional limitations persist despite viral clearance in patients exposed to peg-interferon/ribavirin-containing regimens (ANRS CO13-HEPAVIH cohort). Eur J Gastroenterol Hepatol. 2016 Sep;28(9):1003-7. doi: 10.1097/MEG.0000000000000664. PMID 27177169
- [Result] Marcellin F, Lions C, Rosenthal E, Roux P, Sogni P, Wittkop L, Protopopescu C, Spire B, Salmon-Ceron D, Dabis F, Carrieri MP; HEPAVIH ANRS CO13 Study Group*. No significant effect of cannabis use on the count and percentage of circulating CD4 T-cells in HIV-HCV co-infected patients (ANRS CO13-HEPAVIH French cohort). Drug Alcohol Rev. 2017 Mar;36(2):227-238. doi: 10.1111/dar.12398. Epub 2016 Apr 13. PMID 27073179
- [Result] Carrieri MP, Serfaty L, Vilotitch A, Winnock M, Poizot-Martin I, Loko MA, Lions C, Lascoux-Combe C, Roux P, Salmon-Ceron D, Spire B, Dabis F; ANRS CO13 HEPAVIH Study Group. Cannabis Use and Reduced Risk of Insulin Resistance in HIV-HCV Infected Patients: A Longitudinal Analysis (ANRS CO13 HEPAVIH). Clin Infect Dis. 2015 Jul 1;61(1):40-8. doi: 10.1093/cid/civ217. Epub 2015 Mar 16. PMID 25778750
- [Result] Marcellin F, Roux P, Loko MA, Lions C, Caumont-Prim A, Dabis F, Salmon-Ceron D, Spire B, Carrieri MP; HEPAVIH (ANRS CO13) Study Group. High levels of alcohol consumption increase the risk of advanced hepatic fibrosis in HIV/hepatitis C virus-coinfected patients: a sex-based analysis using transient elastography at enrollment in the HEPAVIH ANRS CO13 cohort. Clin Infect Dis. 2014 Oct 15;59(8):1190-2. doi: 10.1093/cid/ciu525. Epub 2014 Jul 11. No abstract available. PMID 25015913
- [Result] Salmon D, Bani-Sadr F, Gilbert C, Rosenthal E, Valantin MA, Simon A, Neau D, Morlat P, Loko MA, Wittkop L, Dabis F; ANRS CO13HEPAVIH study group. HCV viral load at baseline and at week 4 of telaprevir/boceprevir based triple therapies are associated with virological outcome in HIV/hepatitis C co-infected patients. J Clin Virol. 2015 Dec;73:32-35. doi: 10.1016/j.jcv.2015.10.010. Epub 2015 Oct 19. PMID 26528903
- [Result] ANRS CO13 HEPAVIH Cohort. Regression of liver stiffness after sustained hepatitis C virus (HCV) virological responses among HIV/HCV-coinfected patients. AIDS. 2015 Sep 10;29(14):1821-30. doi: 10.1097/QAD.0000000000000787. PMID 26372388
- [Result] Roux P, Lions C, Cohen J, Winnock M, Salmon-Ceron D, Bani-Sadr F, Sogni P, Spire B, Dabis F, Carrieri MP; ANRS-CO13-HEPAVIH Study Group. Impact of HCV treatment and depressive symptoms on adherence to HAART among HIV-HCV-coinfected patients: results from the ANRS-CO13-HEPAVIH cohort. Antivir Ther. 2014;19(2):171-8. doi: 10.3851/IMP2699. Epub 2013 Oct 28. PMID 24166726
- [Result] Marcellin F, Roux P, Winnock M, Lions C, Dabis F, Salmon-Ceron D, Loko MA, Spire B, Carrieri MP. Using patient-reported outcomes to improve the management of co-infection with HIV and HCV: the ANRS CO13 HEPAVIH cohort. Expert Rev Gastroenterol Hepatol. 2014 May;8(4):351-8. doi: 10.1586/17474124.2014.888949. Epub 2014 Mar 3. PMID 24580042
- [Result] Carrieri MP, Lions C, Sogni P, Winnock M, Roux P, Mora M, Bonnard P, Salmon D, Dabis F, Spire B; ANRS CO13 HEPAVIH Study Group. Association between elevated coffee consumption and daily chocolate intake with normal liver enzymes in HIV-HCV infected individuals: results from the ANRS CO13 HEPAVIH cohort study. J Hepatol. 2014 Jan;60(1):46-53. doi: 10.1016/j.jhep.2013.08.014. Epub 2013 Aug 24. PMID 23978720
- [Result] Bani-Sadr F, Loko MA, Pambrun E, Winnock M, Carrieri P, Gilbert C, Duvivier C, Bouchaud O, Gervais A, Dabis F, Salmon D; ANRS CO 13 HEPAVIH Study Group. Correlates of HIV sustained viral suppression in HIV/hepatitis C virus coinfected patients: possible role of the hepatitis C virus sustained viral response. AIDS. 2014 May 15;28(8):1155-60. doi: 10.1097/QAD.0000000000000218. PMID 24499953
- [Result] Winnock M, Bani-Sadr F, Pambrun E, Loko MA, Carrieri P, Neau D, Morlat P, Marchou B, Dabis F, Salmon D; French National Agency for Research on AIDS and Viral Hepatitis (ANRS) CO13 HEPAVIH Study Group. Factors associated with guideline-based hepatitis C virus (HCV) treatment initiation in HIV/HCV-coinfected patients: role of comorbidities and physicians' perceptions. HIV Med. 2013 Aug;14(7):430-6. doi: 10.1111/hiv.12023. Epub 2013 Mar 5. PMID 23461846
- [Result] Marcellin F, Lions C, Winnock M, Salmon D, Durant J, Spire B, Mora M, Loko MA, Dabis F, Dominguez S, Roux P, Carrieri MP; ANRS CO13 HEPAVIH Study Group. Self-reported alcohol abuse in HIV-HCV co-infected patients: a better predictor of HIV virological rebound than physician's perceptions (HEPAVIH ARNS CO13 cohort). Addiction. 2013 Jul;108(7):1250-8. doi: 10.1111/add.12149. Epub 2013 Mar 21. PMID 23421419
- [Result] Trimoulet P, Merchadou L, Winnock M, Loko MA, Fleury H, Salmon D, Dabis F, Neau D; ANRS CO 13 HEPAVIH Study Group. Hepatitis C virus RNA quantitation in a nationwide French cohort of patients co-infected with HIV and HCV: should the same test be applied to all samples? J Virol Methods. 2012 Apr;181(1):131-3. doi: 10.1016/j.jviromet.2012.01.006. Epub 2012 Jan 20. PMID 22285372
- [Result] Solas C, Pambrun E, Winnock M, Salmon D, Poizot-Martin I, Dominguez S, Bani-Sadr F, Izopet J, Garraffo R, Peytavin G; ANRS CO-13 HEPAVIH Study Group. Ribavirin and abacavir drug interaction in HIV-HCV coinfected patients: fact or fiction? AIDS. 2012 Nov 13;26(17):2193-9. doi: 10.1097/QAD.0b013e32835763a4. PMID 22781224
- [Result] Salmon-Ceron D, Cohen J, Winnock M, Roux P, Sadr FB, Rosenthal E, Martin IP, Loko MA, Mora M, Sogni P, Spire B, Dabis F, Carrieri MP; HEPAVIH group. Engaging HIV-HCV co-infected patients in HCV treatment: the roles played by the prescribing physician and patients' beliefs (ANRS CO13 HEPAVIH cohort, France). BMC Health Serv Res. 2012 Mar 12;12:59. doi: 10.1186/1472-6963-12-59. PMID 22409788
- [Result] Salmon D, Bani-Sadr F, Loko MA, Stitou H, Gervais A, Durant J, Rosenthal E, Quertainmont Y, Barange K, Vittecoq D, Shoai-Tehrani M, Alvarez M, Winnock M, Trinchet JC, Dabis F, Sogni P. Insulin resistance is associated with a higher risk of hepatocellular carcinoma in cirrhotic HIV/HCV-co-infected patients: results from ANRS CO13 HEPAVIH. J Hepatol. 2012 Apr;56(4):862-8. doi: 10.1016/j.jhep.2011.11.009. Epub 2011 Dec 13. PMID 22173166
- [Result] Roux P, Fugon L, Winnock M, Salmon-Ceron D, Lacombe K, Sogni P, Spire B, Dabis F, Carrieri MP; ANRS-CO-13-HEPAVIH Study Group. Positive impact of hepatitis C virus (HCV) treatment on antiretroviral treatment adherence in human immunodeficiency virus-HCV coinfected patients: one more argument for expanded access to HCV treatment for injecting drug users. Addiction. 2012 Jan;107(1):152-9. doi: 10.1111/j.1360-0443.2011.03608.x. Epub 2011 Oct 12. PMID 21819472
- [Result] Loko MA, Bani-Sadr F, Valantin MA, Lascoux-Combe C, Fontaine H, Bonnard P, Gervais A, Bouchaud O, Garipuy D, Quertainmont Y, Vittecoq D, Tehrani MS, Winnock M, Dabis F, Salmon D; ANRS CO 13 HEPAVIH Study Group. Antiretroviral therapy and sustained virological response to HCV therapy are associated with slower liver fibrosis progression in HIV-HCV-coinfected patients: study from the ANRS CO 13 HEPAVIH cohort. Antivir Ther. 2012;17(7):1335-43. doi: 10.3851/IMP2419. Epub 2012 Oct 10. PMID 23052829
- [Result] Carrieri MP, Sogni P, Cohen J, Loko MA, Winnock M, Spire B; HEPAVIH Study Group. Elevated coffee consumption and reduced risk of insulin resistance in HIV-HCV coinfected patients (HEPAVIH ANRS CO-13). Hepatology. 2012 Nov;56(5):2010. doi: 10.1002/hep.25813. No abstract available. PMID 22535683
- [Result] Carrieri MP, Cohen J, Salmon-Ceron D, Winnock M. Coffee consumption and reduced self-reported side effects in HIV-HCV co-infected patients during PEG-IFN and ribavirin treatment: results from ANRS CO13 HEPAVIH. J Hepatol. 2012 Mar;56(3):745-7. doi: 10.1016/j.jhep.2011.08.005. Epub 2011 Aug 31. No abstract available. PMID 21888878
- [Result] Abravanel F, Raymond S, Pambrun E, Winnock M, Bonnard P, Sogni P, Trimoulet P, Dabis F, Salmon-Ceron D, Izopet J; ANRS CO13 HEPAVIH Study Group. HIV-1 tropism and liver fibrosis in HIV-HCV co-infected patients. PLoS One. 2012;7(11):e50289. doi: 10.1371/journal.pone.0050289. Epub 2012 Nov 30. PMID 23226258
- [Result] Winnock M, Bani-Sadr F, Pambrun E, Loko MA, Lascoux-Combe C, Garipuy D, Rosenthal E, Carrieri P, Dabis F, Salmon D. Prevalence of immunity to hepatitis viruses A and B in a large cohort of HIV/HCV-coinfected patients, and factors associated with HAV and HBV vaccination. Vaccine. 2011 Nov 3;29(47):8656-60. doi: 10.1016/j.vaccine.2011.08.125. Epub 2011 Sep 13. PMID 21920402
- [Result] Roux P, Cohen J, Lascoux-Combe C, Sogni P, Winnock M, Salmon-Ceron D, Spire B, Dabis F, Carrieri MP; ANRS-CO13-HEPAVIH study group. Determinants of the underreporting of alcohol consumption by HIV/HCV co-infected patients during face-to-face medical interviews: the role of the physician. Drug Alcohol Depend. 2011 Jul 1;116(1-3):228-32. doi: 10.1016/j.drugalcdep.2010.09.025. Epub 2011 Jan 15. PMID 21239121
- [Result] Loko MA, Bani-Sadr F, Winnock M, Lacombe K, Carrieri P, Neau D, Morlat P, Serfaty L, Dabis F, Salmon D; ANRS CO 13 HEPAVIH Study Group. Impact of HAART exposure and associated lipodystrophy on advanced liver fibrosis in HIV/HCV-coinfected patients. J Viral Hepat. 2011 Jul;18(7):e307-14. doi: 10.1111/j.1365-2893.2010.01417.x. Epub 2011 Jan 11. PMID 21692942
- [Result] Loko MA, Salmon D, Carrieri P, Winnock M, Mora M, Merchadou L, Gillet S, Pambrun E, Delaune J, Valantin MA, Poizot-Martin I, Neau D, Bonnard P, Rosenthal E, Barange K, Morlat P, Lacombe K, Gervais A, Rouges F, See AB, Lascoux-Combe C, Vittecoq D, Goujard C, Duvivier C, Spire B, Izopet J, Sogni P, Serfaty L, Benhamou Y, Bani-Sadr F, Dabis F; ANRS CO 13 HEPAVIH Study Group. The French national prospective cohort of patients co-infected with HIV and HCV (ANRS CO13 HEPAVIH): early findings, 2006-2010. BMC Infect Dis. 2010 Oct 22;10:303. doi: 10.1186/1471-2334-10-303. PMID 20969743
- [Result] Carrieri MP, Cohen J, Winnock M, Salmon D. Chocolate intake, depression, and clinical progression in HIV-HCV coinfected patients: still more questions than answers. Arch Intern Med. 2010 Sep 27;170(17):1607; author reply 1608-9. doi: 10.1001/archinternmed.2010.330. No abstract available. PMID 20876416
- [Result] Cales P, Halfon P, Batisse D, Carrat F, Perre P, Penaranda G, Guyader D, d'Alteroche L, Fouchard-Hubert I, Michelet C, Veillon P, Lambert J, Weiss L, Salmon D, Cacoub P. Comparison of liver fibrosis blood tests developed for HCV with new specific tests in HIV/HCV co-infection. J Hepatol. 2010 Aug;53(2):238-44. doi: 10.1016/j.jhep.2010.03.007. Epub 2010 Apr 18. PMID 20493576
- [Result] Carrieri MP, Protopopescu C, Marcellin F, Rosellini S, Wittkop L, Esterle L, Zucman D, Raffi F, Rosenthal E, Poizot-Martin I, Salmon-Ceron D, Dabis F, Spire B; ANRS CO13 HEPAVIH Study Group. Protective effect of coffee consumption on all-cause mortality of French HIV-HCV co-infected patients. J Hepatol. 2017 Dec;67(6):1157-1167. doi: 10.1016/j.jhep.2017.08.005. Epub 2017 Sep 21. PMID 28942916
- [Result] Yaya I, Roux P, Marcellin F, Salmon-Ceron D, Carrieri MP. Unstable Housing Still a Barrier to Receiving HCV Treatment in France (ANRS CO13 HEPAVIH Cohort). Dig Dis Sci. 2017 Oct;62(10):2943-2944. doi: 10.1007/s10620-017-4703-y. Epub 2017 Aug 5. No abstract available. PMID 28780609
- [Result] Knight R, Roux P, Vilotitch A, Marcellin F, Rosenthal E, Esterle L, Boue F, Rey D, Piroth L, Dominguez S, Sogni P, Salmon-Ceron D, Spire B, Carrieri MP; ANRS CO13-HEPAVIH Study Group. Significant reductions in alcohol use after hepatitis C treatment: results from the ANRS CO13-HEPAVIH cohort. Addiction. 2017 Sep;112(9):1669-1679. doi: 10.1111/add.13851. Epub 2017 Jun 6. PMID 28430385
- [Result] Marcellin F, Protopopescu C, Esterle L, Wittkop L, Piroth L, Aumaitre H, Bouchaud O, Goujard C, Vittecoq D, Dabis F, Salmon-Ceron D, Spire B, Roux P, Carrieri MP; ANRS CO13-HEPAVIH Study Group. Short article: Anger and quality of life in patients co-infected with HIV and hepatitis C virus: a cross-sectional study (ANRS CO13-HEPAVIH). Eur J Gastroenterol Hepatol. 2017 Jul;29(7):786-791. doi: 10.1097/MEG.0000000000000883. PMID 28418984
- [Result] Piroth L, Wittkop L, Lacombe K, Rosenthal E, Gilbert C, Miailhes P, Carrieri P, Chas J, Poizot-Martin I, Gervais A, Dominguez S, Neau D, Zucman D, Billaud E, Morlat P, Aumaitre H, Lascoux-Combe C, Simon A, Bouchaud O, Teicher E, Bani-Sadr F, Alric L, Vittecoq D, Boue F, Duvivier C, Valantin MA, Esterle L, Dabis F, Sogni P, Salmon D; ANRS CO13 HEPAVIH study group. Efficacy and safety of direct-acting antiviral regimens in HIV/HCV-co-infected patients - French ANRS CO13 HEPAVIH cohort. J Hepatol. 2017 Jul;67(1):23-31. doi: 10.1016/j.jhep.2017.02.012. Epub 2017 Feb 22. PMID 28235612
- [Result] Ulveling D, Le Clerc S, Cobat A, Labib T, Noirel J, Laville V, Coulonges C, Carpentier W, Nalpas B, Heim MH, Poynard T, Cerny A, Pol S, Bochud PY, Dabis F, Theodorou I, Levy Y, Salmon D, Abel L, Dominguez S, Zagury JF; HEPAVIH ANRS CO13 Cohort Study Group; Swiss Hepatitis C Cohort Study Group; French ANRS HC EP 26 Genoscan Study Group. A new 3p25 locus is associated with liver fibrosis progression in human immunodeficiency virus/hepatitis C virus-coinfected patients. Hepatology. 2016 Nov;64(5):1462-1472. doi: 10.1002/hep.28695. Epub 2016 Jul 29. PMID 27339598
- [Derived] Chalouni M, Wittkop L, Bani-Sadr F, Lacombe K, Esterle L, Gilbert C, Miailhes P, Zucman D, Valantin MA, Bregigeon-Ronot S, Morlat P, Billaud E, Piroth L, Naqvi A, Sogni P, Salmon D; ANRS CO13 HEPAVIH Cohort Study Group. Risk of severe clinical events after sustained virological response following direct-acting antiviral therapy in HIV and hepatitis C virus coinfected participants. HIV Med. 2021 Oct;22(9):791-804. doi: 10.1111/hiv.13127. Epub 2021 Jul 1. PMID 34212476
- [Derived] Chalouni M, Pol S, Sogni P, Fontaine H, Lacombe K, Marc-Lacombe J, Esterle L, Dorival C, Bourliere M, Bani-Sadr F, de Ledinghen V, Zucman D, Larrey D, Salmon D, Carrat F, Wittkop L; ANRS CO13 HEPAVIH and ANRS CO22 HEPATHER cohort study groups. Increased mortality in HIV/HCV-coinfected compared to HCV-monoinfected patients in the DAA era due to non-liver-related death. J Hepatol. 2021 Jan;74(1):37-47. doi: 10.1016/j.jhep.2020.08.008. Epub 2020 Aug 14. PMID 32798585
- [Derived] Poizot-Martin I, Rosenthal E, Gilbert C, Cano CE, Simon A, Lascoux-Combe C, Alric L, Gervais A, Neau D, Esterle L, Salmon D, Sogni P, Wittkop L; ANRS CO13 HEPAVIH Study Group. Nadir CD4 Is Negatively Associated With Antinuclear Antibody Detection in HCV/HIV-Coinfected Patients. J Acquir Immune Defic Syndr. 2019 Apr 1;80(4):461-466. doi: 10.1097/QAI.0000000000001940. PMID 30570526